CLINICAL TRIAL: NCT03209622
Title: Nicotine Replacement Therapy After Acute Coronary Syndrome
Brief Title: Smoking Cessation After Acute Coronary Syndrome
Acronym: SCACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Sriha Belguith_asma, Head of epidemiology and preventive medicine, Principal Investigator, Associate Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMEMonastir
Record Dates: First submitted 2017-06-20; First posted 2017-07-06 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Smoking; Acute Coronary Syndrome; Recurrence
Keywords: Smoking Cessation; Acute Coronary Syndrome; Cardiology
MeSH Terms: conditions — Smoking; Acute Coronary Syndrome; Recurrence; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Participants hospitalized for acute coronary syndrome were randomly assigned to either group "A", initiating Nicotine replacement therapy (NRT) in intra-hospitalization or a control group "B" that received NRT after hospital discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A intervention (Experimental): intervention = Nicotine replacement therapy (NRT): initiated in cardiology intensive care unit, Some hours after acute coronary syndrome.
  Drug: One or two pachs for each ARM, depending of number of cigarettes consummed every day. The dose is decreased every 4 weeks. The patient leave with an appointment to the external consultation for follow-up.
  Interventions: Procedure: Nicotine replacement therapy delivred in cardiology intensive care unit versus Nicotine replacement therapy delivered after hospital discharge; Drug: Nicotine patch
- B: control (Active Comparator): Intervention: Nicotine replacement therapy (NRT) initiated after hospital discharge, some days after acute coronary syndrome. The patient leave with an appointment to the external consultation for follow-up without pach of nicotine.One or two pachs for each ARM, depending of number of cigarettes consummed every day. The dose is decreased every 4 weeks.
  Interventions: Procedure: Nicotine replacement therapy delivred in cardiology intensive care unit versus Nicotine replacement therapy delivered after hospital discharge; Other: the external consultation

INTERVENTIONS:
Procedure: Nicotine replacement therapy delivred in cardiology intensive care unit versus Nicotine replacement therapy delivered after hospital discharge — when patient is admitted in intensive care of cardiology for acute coronary syndrome he is randomized to Arm A or Arm B
Drug: Nicotine patch — Arm A
  Arms: A intervention
Other: the external consultation — without patch
  Arms: B: control

SUMMARY:
A randomized controlled trial was conducted in cardiology department and smoking cessation center of University Hospital of Monastir (Tunisia). All smokers Hospitalized for ACS were included. Participants were randomly assigned to either group "A", initiating Nicotine replacement therapy (NRT) in intra-hospitalization or a control group "B" that received NRT after hospital discharge. The end point assessment was smoking abstinence at 24 weeks following randomization, defined as self-reported abstinence in the past week before the 24 week clinic visit confirmed by a measured exhaled carbon monoxide ≤8 ppm. Data were analyzed by intention to treat.

DETAILED DESCRIPTION:
Background: Smoking is the main preventable cause worldwide of morbidity and premature death (1). It is a major and independent risk factor for coronary heart disease (CHD) (2). More than two-thirds of sudden cardiac death resulting from acute thrombus occurs in smokers (3). Compared to non-smokers the odds ratio (OR) for myocardial infarction is about 2.5, and for cardiovascular diseases overall the OR is about 2 (2) (4). Smoking cessation in persons with known CHD reduces the risk of recurrent myocardial infarctions or cardiovascular death by 30 % to 50 % (5,6) during the subsequent 3 to 7 years (7). Nevertheless, although smoking cessation is potentially the most effective CHD prevention strategy (5), quitting smoking is difficult and two-thirds of patients will return to smoking within one year of their acute coronary syndrome (ACS) (8,9). So, being hospitalized for a major cardiac condition, such as ACS can be an opportunity to prompt many individuals to stop smoking. Through using this "teachable moment" immediately after an ACS, it may be possible to increase smoking abstinence in this high-risk population (9). Cessation rates among smokers hospitalized for ACS, range from 31% without intervention to 60% with sustained intervention post hospitalization, at one year follow-up (10). Although Nicotine replacement therapy (NRT), Bupropion, and Varenicline have demonstrated efficacy medical treatment for smoking cessation compared with placebo (9). NRT improved cessation rates as well with an OR of 1.84 (95% CI 1.71 to 1.99) (2) and no adverse events was found (1). However, the smoking cessation remains a secondary concern in cardiology departments and there is no well strategies offered to these smoker patients with established CHD. Furthermore, there were no difference in cessation rates between this population and the general population despite the proved benefit of smoking cessation on clinical outcomes in CHD patients (11). Many studies have examined the benefits of smoking cessation after ACS and the efficacy of smoking cessation pharmacotherapy's in hospitalized patients with ACS but few randomized controlled trials have examined the efficacy time of smoking cessation in hospitalized patients with ACS either during the hospitalization or after hospital discharge. We aimed at comparing, among patients with ACS, the smoking cessation rates with NRT when began in-hospitalization, against that began after hospital discharge.

1. Design and study population: We have carried out a randomized controlled trial conducted simultaneously in the smoking cessation center and the department of cardiology at the University Hospital of Monastir (Tunisia). This study was performed from January 2015 to Jun 2016 with a mean of 24 weeks of run-up and 24 weeks of follow-up. We have included patients aged more than 18 years, hospitalized with an ACS actively smoking at the time of inclusion, motivated to quit smoking, able to provide informed consent and willing to participate in a clinical study including a follow-up examination every 2 weeks after hospital discharge. Active smoking was defined as smoking one cigarette or more (or water pipe) per day during the month preceding the hospital stay. Non-inclusion criteria were the refusal of assistance of smoking cessation, inability to follow-up clinical visit (professional, regional or physical hindrance), diagnosis of depression or of serious health condition at admission (ventilated patient, cardiogenic shock, etc).

   Sample size: We hypothesized that nicotine replacement therapy after ACS during hospitalization would improve the rate of smoking cessation rate comparing to that after hospitalization discharge from 32.7% up to 51% . This was considered realistic because of the previous study reported a rate of 51% among smokers who received the NRT in-hospital smoking cessation intervention (12) and 32.7% among patients receiving treatments after hospital discharge (13). The expected sample size of 68 participants would enable us to identify such an increase in the smoking cessation rate with a power of 0.80 and a two-sided p-value of <0.05. The proportion of patients who dropped out or withdrew was expected to be 30%. Hence a sample size of 89 was estimate to be adequate, we have included 99 consecutive patients (14). Computer randomization was performed, after consent was obtained. Blinding was not possible. Participants randomized to arm "A" have received a smoking cessation counseling and a Nicotine Replacement Therapy (NRT) during intra-hospital stay one day after SCA. Those in arm "B" have benefited a smoking cessation counseling during intra-hospital stay, while the NRT was offered on a mean of 14 days after SCA in the first clinical visit after hospital discharge. All patients received a regular follow-up visits in smoking cessation center after hospital discharge every 2 weeks. Of the 99 patients enrolled in the study, 44 (81.4 %) and 30 (66.6 %) patients had respectively completed the follow-up smoking cessation in arm A and arm B. Loss to follow up was equivalent in two arms (p=0.1) (Fig 1).

   Ethical considerations: The study was conducted in accordance with good clinical practice and the ethical standards described in the Helsinki Declaration.
2. Study protocol and data collection:

   During the hospital-stay: All patients included in the two arms study, received an individual therapeutic education associated to motivational interview. The therapeutic education aimed to explain tobacco addiction, psychological, physical and behavioral tobacco dependence, the efficiency of NRT in the smoking cessation and introduce examples of behavioral strategies that the patient might adopt when leaving the hospital to overcome his nicotine dependence. Data was collected through a self-administered questionnaire. Patients were asked about their socio-demographic status, history of tobacco use, level of nicotine dependence (Fagerstrom test for Nicotine Dependence: FTNDs) (15), psychological state (using Hospital Anxiety and Depression Scale (HADS) (16), co-addiction (alcohol, drugs, cannabis) and the level of motivation to quit smoking (QMAT scale) (17). Participants in "A" arm have start NRT. The first appointment was scheduled at one week from hospital discharge.

   After hospital discharge: Participants in "B" arm have start NRT. In the first clinic visit, 2 weeks after SCA event. All patients received a second session of therapeutic education Side effects, symptoms of withdrawal, medication adherence, and smoking status were assessed during follow-up contacts. Smoking status was assessed by self-report of smoking in the preceding 7 days. Self-reported abstinence was confirmed using biochemical validation via exhaled carbon monoxide (ECO) levels. ECO was measured using the CO Check + (18) manufactured by MD Diagnostics Ltd, England. The threshold of exhaled carbon monoxide was a value under 8 ppm. Follow-up involved clinic visits every 2 weeks and phone calls to patients missing their meeting, a new consultation was organized as soon as possible.

   A reduction of NRT dose by a third was required every 28 days and NRT dosage adjustment was done according to signs of under or overdose. During the processing time period, a close collaboration with a team comprised psychiatrists, psychiatrist in addiction and a clinical psychologist to manage the delicate cases such as dual addiction, depression cases and type "A" personalities was required.

   Follow up assessment: The primary end point was 7-day point prevalence smoking abstinence at 24 weeks following randomization, defined as self-reported abstinence in the past week before the 24 week clinic visit confirmed by a measured exhaled carbon monoxide ≤8 ppm. Participants with self-reported abstinence who had exhaled carbon monoxide values >8 ppm, or who reported any smoking in the last week and exhaled carbon monoxide ≤8 ppm were classified as current smokers. Secondary endpoints included measures, by a face-to-face survey, of compliance to medication, the occurrence of side effects of NRT (allergic skin reaction), the withdrawal symptoms (nervousness, headache, lack of concentration, insomnia, and craving) and the benefits of smoking cessation (improvement of respiratory signs, increased appetite, sleep quality improvement, enhancement of physical activity). Compliance to treatment was defined as good if the wearing nicotine patches was on a regular basis.

   End Point Assessment: Smoking cessation status was assessed in 24 weeks visit. Phone survey was performed for patients who have missed their appointments.
3. Statistical analysis Collect and statistical analyses were performed using the SPSS 19.0 statistical software. An initial descriptive analysis involved an examination of the demographic, smoking, and clinical characteristics of the two treatment groups. The primary data analysis examined point prevalence smoking abstinence at 24 weeks. All analyses were intention-to-treat adjusted on the significantly differences between the two arms. Similar to other smoking cessation trials, our analyses assumed that patients who withdrew from the study returned to smoking at their baseline rate. Discrete data are described using proportions, and continuous data are described using means and standard deviations or, in the presence of skewed distributions, medians and interquartile ranges. The data analysis examined point prevalence smoking abstinence at 24 weeks with a comparison between the two treatment groups using 95% CIs based on the binomial distribution. Binary logistic regression was used to determine the factors that were independent predictors of success smoking cessation. Variables included in the multivariate analysis were selected at the significance level of 20 % in the univariate analysis. A p value of 5 % was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 18 years, hospitalized with an ACS actively smoking at the time of inclusion, motivated to quit smoking, able to provide informed consent and willing to participate in a clinical study including a follow-up examination every 2 weeks after hospital discharge.

Exclusion Criteria:

* the refusal of assistance of smoking cessation, inability to follow-up clinical visit (professional, regional or physical hindrance), diagnosis of depression or of serious health condition at admission (ventilated patient, cardiogenic shock, etc).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Smoking is a taboo for Tunisian women especially that live in Monastir, it does not declare their consumptions and the inclusion of the woman can be at the origin of a selection bias
Enrollment: 89 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
smoking cessation rates with NRT among patients hospitalized for acute coronary syndrome | 24 weeks after acute coronary syndrome
  smoking cessation rates with NRT when began in-hospitalization, against that began after hospital discharge

SECONDARY OUTCOMES:
smoking cessation duration with NRT among patients hospitalized for acute coronary syndrome | 24 weeks after acute coronary syndrome
  smoking cessation duration with NRT when began in-hospitalization, against that began after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Elhraiech, A. professor, Study Chair — University hospital of Monastir: Avenue Farhat HACHED 5000 Monastir Tunisia; Asma Sriha Belguith, Professor, Principal Investigator — University hospital of Monastir: Avenue Farhat HACHED 5000 Monastir Tunisia
Locations (1):
- Abroug, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
individual participant data have been invited and study results have been presented

REFERENCES:
- [Background] Cahill K, Lindson-Hawley N, Thomas KH, Fanshawe TR, Lancaster T. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2016 May 9;2016(5):CD006103. doi: 10.1002/14651858.CD006103.pub7. PMID 27158893
- [Background] Barth J, Jacob T, Daha I, Critchley JA. Psychosocial interventions for smoking cessation in patients with coronary heart disease. Cochrane Database Syst Rev. 2015 Jul 6;2015(7):CD006886. doi: 10.1002/14651858.CD006886.pub2. PMID 26148115
- [Background] Yahagi K, Joner M, Virmani R. Impact of smoking on coronary heart disease: is there a smoker's paradox? Coron Artery Dis. 2015 Sep;26(6):466-8. doi: 10.1097/MCA.0000000000000274. No abstract available. PMID 26217891
- [Background] Baccouche H, Belguith AS, Boubaker H, Grissa MH, Bouida W, Beltaief K, Sekma A, Fredj N, Bzeouich N, Zina Z, Boukef R, Soltani M, Nouira S. Acute coronary syndrome among patients with chest pain: Prevalence, incidence and risk factors. Int J Cardiol. 2016 Jul 1;214:531-5. doi: 10.1016/j.ijcard.2015.11.065. Epub 2015 Nov 11. PMID 26586217
- [Background] Holtrop JS, Stommel M, Corser W, Holmes-Rovner M. Predictors of smoking cessation and relapse after hospitalization for acute coronary syndrome. J Hosp Med. 2009 Mar;4(3):E3-9. doi: 10.1002/jhm.415. PMID 19301384
- [Background] Chow CK, Jolly S, Rao-Melacini P, Fox KA, Anand SS, Yusuf S. Association of diet, exercise, and smoking modification with risk of early cardiovascular events after acute coronary syndromes. Circulation. 2010 Feb 16;121(6):750-8. doi: 10.1161/CIRCULATIONAHA.109.891523. Epub 2010 Feb 1. PMID 20124123
- [Background] Windle SB, Bata I, Madan M, Abramson BL, Eisenberg MJ. A randomized controlled trial of the efficacy and safety of varenicline for smoking cessation after acute coronary syndrome: design and methods of the Evaluation of Varenicline in Smoking Cessation for Patients Post-Acute Coronary Syndrome trial. Am Heart J. 2015 Oct;170(4):635-640.e1. doi: 10.1016/j.ahj.2015.07.010. Epub 2015 Jul 17. PMID 26386786